CLINICAL TRIAL: NCT06029062
Title: tACS Brain Neuromodulation for Sensory and Motor Recovery After Neurological Impairments
Brief Title: tACS for Sensory Motor Recovery After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sheng Li, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-22-0046 (Experiment 1)
Record Dates: First submitted 2023-05-10; First posted 2023-09-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Motor Recovery
Keywords: tACS; Motor recovery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- tACS Sham, tACS 10Hz, tACS 20Hz (Experimental): tACS Sham is a temporary non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for up to 30 second, it is not designed to entrain neuronal activity into any external regulatory frequency patterns.
  tACS 10Hz is a 10Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp or 20 or 40 minutes to entrain neuronal activity into 10Hz frequency patterns.
  tACS 20Hz is a 20Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for 20 or 40 minutes to entrain neuronal activity into 20Hz frequency patterns.
  Interventions: Device: tACS Sham; Device: tACS 10Hz; Device: tACS 20Hz
- HD-tACS 20Hz, HD-tACS 10Hz, HD-tACS Sham (Experimental): tACS Sham is a temporary non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for up to 30 second, it is not designed to entrain neuronal activity into any external regulatory frequency patterns.
  tACS 10Hz is a 10Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp or 20 or 40 minutes to entrain neuronal activity into 10Hz frequency patterns.
  tACS 20Hz is a 20Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for 20 or 40 minutes to entrain neuronal activity into 20Hz frequency patterns.
  Interventions: Device: tACS Sham; Device: tACS 10Hz; Device: tACS 20Hz
- HD-tACS 10Hz, HD-tACS 20Hz, HD-tACS Sham (Experimental): tACS Sham is a temporary non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for up to 30 second, it is not designed to entrain neuronal activity into any external regulatory frequency patterns.
  tACS 10Hz is a 10Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp or 20 or 40 minutes to entrain neuronal activity into 10Hz frequency patterns.
  tACS 20Hz is a 20Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for 20 or 40 minutes to entrain neuronal activity into 20Hz frequency patterns.
  Interventions: Device: tACS Sham; Device: tACS 10Hz; Device: tACS 20Hz

INTERVENTIONS:
Device: tACS Sham — Sham tACS will applied to the brain through the scalp for 20 minutes.
Device: tACS 10Hz — 10Hz tACS will applied to the brain through the scalp for 20 minutes.
Device: tACS 20Hz — 20Hz tACS will applied to the brain through the scalp for 20 minutes.

SUMMARY:
The overall goal is to investigate the effectiveness of a novel intervention - transcranial alternating current stimulation (tACS) for motor recovery in stroke survivors.

ELIGIBILITY:
Inclusion/exclusion criteria for stroke subjects

Inclusion criteria:

1. Age between 18~75 years old
2. ≥ 6 months post stroke, medically stable;
3. Unilateral, single stroke (no restriction on type (ischemic or hemorrhagic) or volume (large or small) of stroke);
4. Visible finger flexor activation/movement
5. The ability to give consent

Exclusion criteria:

1. Patients with visual deficit/neglect; hearing or cognitive impairment;
2. Patients that are currently adjusting tone alternating medications (e.g., baclofen), or
3. Patients received botulinum toxin injection to the arm/fingers <4 months, or phenol injections <2 years;
4. Patients with pacemaker, metal implants or supplemental oxygen;
5. Patients who have musculoskeletal disorders, including pain in the affected side
6. Women who are pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Block and Box Test (BBT) of Motor functional test | Change of BBT performance 5 minutes before and 5 minutes after the tACS intervention will be measured.
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick and simple test used with a wide range of populations, including clients with stroke.
EEG alpha band and Beta band | Change of EEG alpha band and Beta band 5 minutes before and 5 minutes after the tACS intervention will be measured.
  Electroencephalography (EEG) is valuable to infer and evaluate the neural interaction. Components of the alpha and beta frequency bands like the sensorimotor rhythm originated from the primary motor cortex and related brain areas reflect human movement. The power of 8-13 Hz alpha and 14-30 Hz beta frequency bands will be used for the classification.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Li, MD, Ph.D, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No